CLINICAL TRIAL: NCT00708747
Title: Biseko Versus Albumin in the Treatment of High Risk Patients With Systemic Inflammatory Response Syndrome - a Randomized Controlled Trial
Brief Title: Biseko Versus Albumin in Systemic Inflammatory Response Syndrome (SIRS) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Frass, Medical University Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2340
Record Dates: First submitted 2008-06-26; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-07

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Immunoglobulins; inhibitor proteins; human albumin; systemic inflammatory response syndrome; interleukins; standardized serum-protein solution
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): Patients were randomised to receive a commercially available standardised 5% serum-protein solution (Biseko, Biotest, Dreieich, Germany) containing all important transport and inhibitor proteins as well as immunoglobulins
  Interventions: Drug: Biseko
- A (Active Comparator): Patients were randomised to receive a 5% albumin solution
  Interventions: Drug: Albumin (5% serum-protein solution containing immunoglobulins)

INTERVENTIONS:
Drug: Albumin (5% serum-protein solution containing immunoglobulins) — 5% albumin was given intravenously at a volume of 1,000 ml on the first day and 500 ml/day during the following four days.
  Other Names: Albumin
  Arms: A
Drug: Biseko — Standardised 5% serum-protein solution (Biseko, Biotest, Dreieich, Germany) was given intravenously at a volume of 1,000 ml on the first day and 500 ml/day during the following four days.
  Arms: B

SUMMARY:
Morbidity and mortality in patients suffering from systemic inflammatory response syndrome (SIRS) remain high. The primary aim of the present study is to assess the efficacy of a standardized 5% serum-protein solution containing immunoglobulins on serum cytokine levels. The secondary aim is to evaluate survival of the patients.

DETAILED DESCRIPTION:
Out of 40 patients randomised, 18 patients received albumin, 20 patients received Biseko and 2 patients died before receiving the complete study medication. During days 1-6 of the study period, serum-levels of IL-1ß were significantly lower in patients with Biseko-therapy compared to patients receiving albumin (IL-1ß-Area under the curve 65.04 ± 71.09 days.pg/ml and 111.05 ± 156.97 days.pg/ml respectively, P=0.03). No difference could be found in serum-levels of IL-6, TNF-α and TNF-R between both groups. While a statistically not significant trend towards better survival was observed in the Biseko-group on day 28, the survival rate on day 180 was significantly higher in the Biseko-group [9/18 (50%)] vs. albumin- group [2/20 (10%), (P=0.008)].

Conclusion: Data suggest that Biseko treatment was associated with significantly lower IL-1ß plasma concentrations (d1 to 6) and improved long-term survival rates.

The data provided in our study are the first to be collected in a randomized, controlled trial. Certainly, the small number of patients and the variety of diseases limit our study, however, the variety of diseases reflects the realistic large scale of morbidity in the medical intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85 years fulfilling at least two of the four SIRS criteria:

  * body temperature > 38°C or < 36°C
  * tachycardia > 90/min
  * tachypnea > 20/min with spontaneous respiration
  * leucocytosis > 12,000/mcl
  * leucopenia < 4,000/mcl or more than 10 % immature granulocytes were included [8,21,22]

Exclusion Criteria:

* Patients with proven intolerance against homologous protein solutions
* Patients with known liver failure
* Pregnant patients
* Patients with absolute IgA deficiency were excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-07; Primary Completion 2001-06 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
The primary aim of the present study is to assess the efficacy of a standardized 5% serum-protein solution containing immunoglobulins on serum cytokine levels. | 3 years

SECONDARY OUTCOMES:
The secondary aim is to evaluate survival of the patients. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

REFERENCES:
- [Background] Vincent JL, Gerlach H. Fluid resuscitation in severe sepsis and septic shock: an evidence-based review. Crit Care Med. 2004 Nov;32(11 Suppl):S451-4. doi: 10.1097/01.ccm.0000142984.44321.a4. PMID 15542955